CLINICAL TRIAL: NCT00919217
Title: Exploratory Study on the Timing of MS Symptoms
Brief Title: Exploratory Study on the Timing of Multiple Sclerosis (MS) Symptoms
Status: Recruiting | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Cynthia Corbitt, Associate Professor, University of Louisville
Other Study IDs: 08.0172
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Relapsing-remitting multiple sclerosis; RR-MS; Women
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Relapsing-remitting multiple sclerosis: Females with relapsing-remitting multiple sclerosis

SUMMARY:
The investigators' overall hypothesis is that appearance or worsening of relapsing-remitting multiple sclerosis (RR-MS) symptoms are affected by various factors including stress, hormonal cycles, illness and missed medications.

DETAILED DESCRIPTION:
Fluctuations in MS symptoms in women with RR-MS might be affected by a variety of factors. To determine which factors are important, we are asking subjects to fill out a diary and calendar on a daily basis for 90 days. After an initial instructional meeting over the phone, the materials are filled out at home and returned monthly via postage-paid envelopes provided by the study. Compensation ($10 gift card) is sent after each monthly diary is received. The diary includes a list of symptoms and a rank scale for the women to show subtle changes in MS symptoms. The calendar allows the subject to denote additional factors such as stress, hormonal cycles, illnesses or immunizations and changed or missed medications. We anticipate that statistical analysis will reveal which of these factors affect women with relapsing-remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* females
* diagnosed with relapsing-remitting multiple sclerosis

Exclusion Criteria:

* male
* no diagnosis of relapsing-remitting MS
* diagnosis of any other autoimmune disease or fibromyalgia
* peri-, post-, or surgically menopausal
* pregnant within past year or nursing
* history of chemotherapy
* on experimental medications
* treatment with steroids in the last 30 days

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females with relapsing-remitting multiple sclerosis, not menopausal, neither pregnant nor nursing, not treated with steroids in the last 30 days and not on experimental medications
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
number of days with appearance or worsening of symptoms | 3 months

SECONDARY OUTCOMES:
timing of appearance or worsening of symptoms | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Corbitt, PhD, Principal Investigator — University of Louisville, Dept. Biology
Locations (1):
- University of Louisville (recruiting nationwide), Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided